CLINICAL TRIAL: NCT00838240
Title: Clofarabine in Combination With a Standard Remission Induction Regimen (AraC and Idarubicin) in Patients 18-60 Years Old With Previously Untreated Intermediate and Bad Risk Acute Myelogenous Leukemia (AML) or High Risk Myelodysplasia (MDS) : a Phase I-II Study of the EORTC-LG and GIMEMA (AML-14A Trial)
Brief Title: Clofarabine, Cytarabine, and Idarubicin in Treating Patients With Intermediate-Risk or High-Risk Acute Myeloid Leukemia or High-Risk Myelodysplasia
Acronym: AML-14A
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-06061; EORTC-06061; EU-20905; 2006-004912-28 (EudraCT Number); GIMEMA-AML-14A
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with inv(16)(p13;q22); untreated adult acute myeloid leukemia; de novo myelodysplastic syndromes; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities | interventions — Clofarabine; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive idarubicin IV over 5 minutes on days 1, 3, and 5, cytarabine IV continuously on days 1-10, and clofarabine IV over 1 hour on days 2, 4, 6, 8, and 10.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: idarubicin
- Arm II (Experimental): Patients receive idarubicin IV and cytarabine IV as in arm I. Patients also receive clofarabine IV by push injection over 10 minutes on days 2, 4, 6, 8, and 10.
  Interventions: Drug: clofarabine; Drug: cytarabine; Drug: idarubicin

INTERVENTIONS:
Drug: clofarabine — Given IV
Drug: cytarabine — Given IV
Drug: idarubicin — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, cytarabine, and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of clofarabine and to see how well it works when given together with cytarabine and idarubicin in treating patients with intermediate-risk or high-risk acute myeloid leukemia or high-risk myelodysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the optimum dose of clofarabine in combination with cytarabine and idarubicin in patients with previously untreated intermediate- and high-risk acute myeloid leukemia or high-risk myelodysplasia. (Phase I)
* To determine the safety and tolerance of this regimen in order to determine the recommended phase II dose. (Phase I)
* To explore the antitumor activity of this regimen in these patients. (Phase II)
* To determine the activity expressed as complete remission (CR)/CR with incomplete hematopoietic recovery (CRi) rate following induction therapy. (Phase II)

Secondary

* To determine the activity expressed as CR/CRi rate following induction (1 or 2 courses) and consolidation therapy. (Phase I)
* To determine hematopoietic recovery (platelets and neutrophils) after induction and consolidation therapy.
* To determine safety and tolerability of this regimen. (Phase II)
* To determine activity expressed as CR/CRi rate after consolidation therapy. (Phase II)
* To determine feasibility of blood CD34 harvesting after consolidation therapy. (Phase II)
* To determine disease-free and overall survival from CR/CRi. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of clofarabine followed by an randomized phase II study. Patients are stratified according to center, and presence of poor prognostic features (WBC at diagnosis ≥ 100,000/μL vs presence of very high risk cytogenetic features -5/5q-, -7/7q-, presence of complex abnormalities [> 3 abnormalities], 3q, t[6;9], or t[9;22]). Patients are randomized to 1 of 2 treatment arms.

* Induction therapy:

  * Arm I: Patients receive idarubicin IV over 5 minutes on days 1, 3, and 5, cytarabine IV continuously on days 1-10, and clofarabine IV over 1 hour on days 2, 4, 6, 8, and 10.
  * Arm II: Patients receive idarubicin IV and cytarabine IV as in arm I. Patients also receive clofarabine IV by push injection over 10 minutes on days 2, 4, 6, 8, and 10.
* Consolidation therapy: Patients receive cytarabine IV over 2 hours every 12 hours on days 1-6 and idarubicin IV over 5 minutes once daily on days 4-6.

After completion of study therapy, patients are followed periodically for 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following by WHO criteria:

  * Acute myeloid leukemia (AML) (≥ 20% bone marrow blasts by bone marrow aspiration or biopsy)

    * No acute promyelocytic leukemia (M3)
    * All cytogenetic groups allowed, except for the following:

      * t(15;17)
      * t(8;21) or inv(16) AND a WBC count at diagnosis of < 100,000/μL
    * Primary or secondary AML allowed, including AML after myelodysplasia (MDS)
  * High-risk MDS (≥ 10% bone marrow blasts by bone marrow aspiration or biopsy)
* No chronic myelogenous leukemia in blast crisis or AML supervening a myeloproliferative disorder
* Previously untreated disease, except for ≤ 14 days of hydroxyurea
* No CNS leukemia

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Serum creatinine ≤ 1.0 mg/dL or glomerular filtration rate > 60 mL/min
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* ALP ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for ≥ 3 months after completion of study treatment
* No active uncontrolled infection
* No HIV positivity
* No psychological, familial, sociological, or geographical conditions precluding compliance with study treatment or follow up
* No concurrent severe uncontrolled cardiovascular disease (i.e., symptomatic congestive heart failure or symptomatic ischemic heart disease [NYHA class III-IV])
* No concurrent malignant disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent cytotoxic drugs or experimental therapies (e.g., antiangiogenic drugs, tyrosine kinase inhibitors)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity as assessed by CTCAE v3.0 (Phase I)
Response rate (Phase II)

SECONDARY OUTCOMES:
Toxicity as assessed by CTCAE v3.0 (Phase II)
Response rate (Phase I)
Duration of survival
Duration of survival from complete remission (CR)/CR with incomplete hematopoietic recovery (CRi) rate
Disease-free survival from CR/CRi
Incidence of relapse and incidence of death in CR/CRi

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, Principal Investigator — EORTC (Phase I) - Leiden University Medical Center, NL; Dominik Selleslag, Principal Investigator — EORTC (Phase II) - AZ Sint-Jan, BE; Giovanna Meloni, Principal Investigator — GIMEMA (Phase I & II) - Universita Degli Studi "La Sapienza", IT
Locations (10):
- Belgium (3):
  - A.Z. Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - CHU Sart-Tilman, Liège
- University Hospital Rebro, Zagreb, Croatia
- Hôpital Saint Antoine AP-HP, Paris, France
- Italy (2):
  - Azienda Ospedallera Universitaria - Policlinico Tor Vergata, Roma
  - Univesita Degli Studi "La Sapienza", Roma
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Leiden University Medical Center, Leiden
  - Radboud University Nijmegen Medical Center, Nijmegen